CLINICAL TRIAL: NCT05048017
Title: Regorafenib Combined With PD-1 Inhibitor Therapy for Second-line Treatment of Hepatocellular Carcinoma: A Single Arm, Nonrandomized, Single Center Clinical Study
Brief Title: Regorafenib Combined With PD-1 Inhibitor Therapy for Second-line Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-3039
Record Dates: First submitted 2021-08-17; First posted 2021-09-17 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma; Regorafenib; PD-1 Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib; Immune Checkpoint Inhibitors; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regorafenib plus PD-1 inhibitor (Experimental): Regorafenib (BAY 73-4506, Stivarga®) is an oral diphenylurea multi-kinase inhibitor that targets angiogenic (VEGFR1-3, TIE2), stromal (PDGFR-β, FGFR), and oncogenic receptor tyrosine kinases (KIT, RET, and RAF).
  Camrelizumab (AiRuiKa™), a programmed cell death 1 (PD-1) inhibitor being developed by Jiangsu Hengrui Medicine Co. Ltd, recently received conditional approval in China for the treatment of relapsed or refractory classical Hodgkin lymphoma.
  Toripalimab, a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2), is being developed by Shanghai Junshi Bioscience Co., Ltd in China for the treatment of various cancers.
  Pembrolizumab (Keytruda) the programmed cell death protein 1 (PD1) is one of the checkpoints that regulates the immune response. Ligation of PD1 with its ligands PDL1 and PDL2 results in transduction of negative signals to T-cells.
  Interventions: Drug: Regorafenib; Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: Regorafenib — Regorafenib, 120 mg, once a day, 3 weeks on/1 week off
  Other Names: BAY 73-4506, Stivarga
Drug: PD-1 inhibitor — Camrelizumab: 200mg (BW ≥ 50 kg) or 3 mg/kg (BW < 50 kg) Toripalimab: 240mg is given through intravenous drip every 3 weeks on Day 1 of each course of treatment.
  Pembrolizumab: 200mg is given through intravenous drip every 3 weeks.
  Other Names: Camrelizumab (AiRuiKa™)、Toripalimab、Pembrolizumab(Keytruda)

SUMMARY:
This is a single arm, nonrandomized, single center clinical study to investigate the safety and efficacy of regorafenib combined with PD-1 inhibitor therapy for second-line treatment of hepatocellular carcinoma

DETAILED DESCRIPTION:
To observe and evaluate the efficacy, safety and biomarker analysis of regorafenib combined with PD-1 inhibitor for the second-line treatment of hepatocellular carcinoma.In this study, 20 patients with hepatocellular carcinoma will be enrolled for regorafenib combined with PD-1 inhibitor therapy.In the absence of any of the following conditions, such as withdrawal of informed consent by subjects, intolerable drug side effects, or the investigator's determination that further study is not appropriate, the expected study treatment for each subject will continue until radiologically confirmed tumor progression. Efficacy indicators and safety indicators will be observed during the trial.

ELIGIBILITY:
Inclusion criteria

Subject must meet all of the following criteria to be enrolled in the study:

1. Subjects volunteer to participate in the study, agree to sign their written informed consent, show good compliance and are cooperative with the follow-up.
2. There is no gender requirement but age requirement (age>18) for the subjects who sign the informed consent.
3. The subjects were diagnosed as advanced hepatocellular carcinoma (HCC) by imaging or histological examination.
4. The disease is not suitable for radical surgery and/or local treatment, or disease progression occurs after surgery and/or local treatment.
5. The patients with at least one measurable lesion according to RECIST, version1.1, and no local radiotherapy was performed. Results of spiral CT scan (RECIST, version 1.1): LD (lesion) ≥ 10 mm or SD (enlarged lymph node) ≥ 15 mm.
6. The patients who failed or were intolerable to the following treatments: simple sorafenib therapy, or sorafenib combined with PD-1 therapy, or simple lenvatinib therapy, or lenvatinib combined with PD-1 therapy, or bevacizumab combined with atezolizumab.
7. Definition of treatment failure: It refers to the disease progression during treatment or the recurrence of the disease after treatment (Obvious disease recurrences and progressions appeared in patients who have received at least one radical or palliative resection, interventional therapy or radiotherapy. The treatment period of systemic chemotherapy like oxaliplatin and other systemic chemotherapy must be at least one cycle. The treatment time of molecular targeted therapy must be longer than 14 days).
8. Definition of intolerable: Hematological toxicity ≥ Grade IV, or non-hematological toxicity ≥ Grade III, or damage to the heart, liver, kidney and other major organs ≥ Grade II occurred during the treatment. For details, please refer to the package inserts of each drug.
9. The ECOG score within 1 week before enrollment was 0-1 points.
10. Child-Pugh score for liver function: Class A, BCLC staging is B-C stage.
11. The time from failure of first-line system treatment to enrollment in this study (the time to sign the informed consent form) was ≥ 2 weeks , and the adverse events basically returned to normal (NCI-CTCAE ≤ Grade I).
12. The expected survival time is greater than or equal to 6 months.
13. HBV DNA < 2000 IU/ml (104 copies/ml).
14. Hematology and organ function are adequate, based on the following laboratory test results obtained within 14 days prior to the start of study treatment (unless otherwise stated):

    14.1 Routine blood test: (No blood transfusion, G-CSF treatment, or medication correction within 14 days prior to screening) 14.2 Hb ≥ 100 g/L; Neutrophils ≥ 1.5 × 109/L; PLT ≥ 75 × 109/L 14.3 Biochemical examination: (No ALB was administered within 14 days) ALB ≥ 35 g/L; ALT and AST<3×ULN; TBIL ≤ 2×ULN; Creatinine ≤ 1.5×ULN; PT ≤ ULN+4S; INR ≤ 2.2 (In the Child-Pugh score, only one of albumin and bilirubin can be scored as 2 points)
15. No active autoimmune disease requiring systemic treatment in the past 2 years (i.e. using disease modulators, corticosteroids, or immunosuppressive agents). Alternative therapy (e.g., physiological corticosteroid replacement therapy for thyroxine, insulin, or adrenal or pituitary insufficiency, etc.) is not considered as a form of systemic therapy.
16. Reproductive women: Agree to abstain from sex (avoid heterosexual intercourse) or use a contraceptive method with an annual contraceptive failure rate < 1% during treatment and for at least 6 months after the last administration.

    16.1 If the female patient has menstruation and has not yet reached the post-menopausal state (continuous non-menstrual period ≥ 12 months, with no other reasons other than menopause are found), and have not undergone sterilization (removal of the ovaries and/or uterus), it is considered that the patient is fertile.

    16.2 Examples of contraceptive methods with an annual contraceptive failure rate < 1% include bilateral fallopian tube ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper-ring intrauterine devices.

    16.3 The reliability of sexual control should be evaluated relative to the duration of the clinical trial and the preferred and daily lifestyle of the patient. Periodic abstinence (for example, calendar days, ovulatory period, symptomatic body temperature, or post-ovulation methods) and external ejaculation are unacceptable methods of contraception.
17. Male: Agree to abstinence (not having heterosexual intercourse) or use contraceptive measures, and agree not to donate sperm, defined as follows:

    17.1 When his female partner has fertility, the male patient must abstain from sex during treatment and within 6 months after the last administration, or use condoms and other contraceptive methods to make the annual contraceptive failure rate < 1%. Male patients must agree not to donate sperm during the same time period. When his female partner is pregnant, the male patient must abstain from sex or use a condom for contraception during the treatment period and within 6 months after the last dose to avoid the fetus being affected by the study.
18. The reliability of sexual control should be evaluated relative to the duration of the clinical trial and the preferred and daily lifestyle of the patient. Periodic abstinence (for example, calendar days, ovulatory period, symptomatic body temperature, or post-ovulation methods) and external ejaculation are unacceptable methods of contraception.
19. Before the first dose of study medication for biomarker analysis, archived tumor tissue or new tissue biopsy specimens must be available. In the case when the archived tissue cannot be provided, and the biopsy cannot be performed, participants can consult the investigator and join the group after obtaining the investigator's consent.

Note: If an unstained section is submitted, the new section should be submitted to the testing laboratory within 14 days after cutting.

Exclusion criteria：

Patients meeting one or more of the following conditions cannot be included:

1. The clinical stage is stage IV, and/or patients with hepatobiliary solid tumors with any of the following conditions:

   1.1 The patient is suitable for surgical radical treatment, 1.2 or, the patient has accepted radical treatment and has no assessable lesion, 1.3 or, the patient has a history of liver transplantation or plans to undergo liver transplantation.
2. Patient who is known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components; Patient who is known to be allergic to regorafenib and its components.
3. ECOG score ≥ 2 points.
4. Patient who has ascites with clinical symptoms, that requires therapeutic abdominal puncture or drainage, or Child-Pugh score > 2 points.
5. Patient with serious heart, cerebrovascular and other systemic diseases with unstable or uncontrollable condition.
6. Patient with active central nervous system (CNS) metastasis and/or cancerous meningitis. Subjects with previously treated brain metastases can participate in the study, as long as their brain metastases are stable (imaging shows no evidence of progression for at least four weeks before the first trial treatment and all neurological symptoms have returned to baseline) with no evidence shows new or enlarged brain metastases, and steroids are not used for at least 7 days before the trial treatment. This exception does not include cancerous meningitis, which is excluded regardless of how its clinical stability is.
7. Patient who has accepted major surgery within 4 weeks before the first study administration (appropriate wound healing and clinical evaluation must be performed after major surgery, which has nothing to do with the time of enrollment)
8. Patient with liver and kidney dysfunction, such as jaundice, ascites, and/or bilirubin > 2×ULN, and/or alkaline phosphatase ≥ 3×ULN; and/or ≥ Grade 3 (CTC-AE 5.0) persistent proteinuria, creatinine ratio > 3.5g/24 hours, or renal failure requiring blood or peritoneal dialysis, etc.
9. Urine routine test shows urine protein ≥ ++ or confirmed 24-hour urine protein quantification>1.0g;
10. Patient with persistent infection which is greater than Grade 2 (CTC-AE5.0).
11. Patient with a history of organ allogeneic transplantation (participants underwent allogeneic tissue/solid organ transplantation)
12. Patient with a history of active tuberculosis (TB bacilli)
13. Patient intolerance to any study drug (or any excipient)
14. Female patient who is pregnant, breastfeeding, or who does not accept contraceptive measures.
15. Patient with known or untreated brain metastases, or with epilepsy which needs medication.
16. Patient with bone metastases who have received palliative radiotherapy (radiotherapy area > 5% bone marrow area) within 4 weeks before participating in the study, or patient who has unhealed wounds, ulcers or fractures, or has a history of organ transplantation.
17. Patient with a history of gastrointestinal bleeding or a clear gastrointestinal bleeding tendency within the past 6 months, such as: esophageal varices with bleeding risk, local active ulcer lesions and fecal occult blood ≥ (++). Gastroscopy is needed for patients with stool occult blood (+);
18. There is evidence or history of bleeding mechanism disorders such as bleeding events ≥ Grade 3 (CTC-AE5.0).
19. Patient with a history of human immunodeficiency virus (HIV) infection.
20. Patient who tests positive for hepatitis B or C and has not received regular treatment.
21. Patient with severe non-healing wounds, ulcers or fractures
22. Patient treated with regorafenib beforehand.
23. Patient diagnosed of immunodeficiency or received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment. After consultation with the sponsor, the use of physiological doses of corticosteroids (not exceeding 7.5 mg/d prednisone or equivalent doses of similar drugs) can be approved.
24. Existence of drug abuse; or any medical, psychological or social condition that may affect the research and patient compliance, or even endanger patient safety.
25. There are many factors that affect oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction, and conditions which significantly affect the administration and absorption of drugs).
26. There is unresolved toxicity > Grade 1 caused by any previous treatment/manipulation (CTC-AE5.0, except for hair loss, anemia, and hypothyroidism).
27. Patient who received live virus vaccine within 30 days of the planned start of treatment. Seasonal influenza vaccine without live virus is allowed.
28. Patients with objective evidence showing pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired lung function, etc. in the past and at present.
29. Patient who received strong CYP3A4 inhibitor treatment within 7 days before participating in the study, or received strong CYP3A4 inducer treatment within 12 days before participating in the study.
30. Patient who is participating in another clinical study at the same time.
31. Patient who was considered to be unsuitable to participate in this study after the investigator comprehensively judged the condition.

Termination criteria：

1. The subject withdraws the informed consent and asks to withdraw.
2. Medical imaging examination confirms the progression of disease, and the treatment is not beneficial for disease progression through clinical judgment.
3. After dose adjustment, the subject still cannot tolerate toxicity.
4. Other conditions that the investigator considers necessary for the subject to withdraw from the study.
5. The sponsor terminates the study due to security concerns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | one year
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1) or death of any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients
Complete response (CR) | one year
  Disappearance of all target lesions, no appearance of new lesions, and normalization of tumor markers last for at least 4 weeks.
Partial response (PR) | one year
  Sum of the maximum diameters of target lesions is reduced by at least 30%, which lasts for at least 4 weeks.
Overall survival (OS) | one year
  It is the time from when a subject is clearly enrolled to death from any cause.
Duration of response (DOR) | one year
  It is the time from the first-time PR or CR (subject to the earlier one) objectively reported to the first-time disease progression or death.
Percentage of patients with stable disease (SD) ≥ 4 weeks | one year
  It is specifically referred to the percentage of patients with identified SD that can be evaluated for efficacy.
Progression-free survival rate at 3 months | 6 months
  It's the percentage of patients with no disease progression or died from any cause after 3 months of treatment with combination of regorafenib and PD-1 inhibitor in the total number of patients whose efficacy can be evaluated.
Mortality at 12 months | one year and a half
  It's the percentage of patients who died of any cause after 12 months treatment with combination of regorafenib and PD-1 inhibitor in total enrolled patients.

OTHER OUTCOMES:
Adverse Event (AE) | two years
  Definition: Refers to any adverse medical event that occurs in patients receiving medical product treatment or subjects of clinical studies, which may not have a causal relationship with the treatment. AE includes but is not limited to: abnormal laboratory test results; clinically significant symptoms and signs; allergies, etc.
Adverse Drug Reaction (ADR) | two years
  All noxious and unintended responses to a medicinal product related to any dose should be considered adverse drug reactions. The phrase "responses to a medicinal products" means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility, i.e., the relationship cannot be ruled out.

CONTACTS AND LOCATIONS:
Locations (1):
- Hai-Tao Zhao, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Background] Kamangar F, Dores GM, Anderson WF. Patterns of cancer incidence, mortality, and prevalence across five continents: defining priorities to reduce cancer disparities in different geographic regions of the world. J Clin Oncol. 2006 May 10;24(14):2137-50. doi: 10.1200/JCO.2005.05.2308. PMID 16682732
- [Background] Richman DM, Tirumani SH, Hornick JL, Fuchs CS, Howard S, Krajewski K, Ramaiya N, Rosenthal M. Beyond gastric adenocarcinoma: Multimodality assessment of common and uncommon gastric neoplasms. Abdom Radiol (NY). 2017 Jan;42(1):124-140. doi: 10.1007/s00261-016-0901-x. PMID 27645897
- [Background] Ryerson AB, Eheman CR, Altekruse SF, Ward JW, Jemal A, Sherman RL, Henley SJ, Holtzman D, Lake A, Noone AM, Anderson RN, Ma J, Ly KN, Cronin KA, Penberthy L, Kohler BA. Annual Report to the Nation on the Status of Cancer, 1975-2012, featuring the increasing incidence of liver cancer. Cancer. 2016 May 1;122(9):1312-37. doi: 10.1002/cncr.29936. Epub 2016 Mar 9. PMID 26959385
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Background] Qin S, Ren Z, Meng Z, Chen Z, Chai X, Xiong J, Bai Y, Yang L, Zhu H, Fang W, Lin X, Chen X, Li E, Wang L, Chen C, Zou J. Camrelizumab in patients with previously treated advanced hepatocellular carcinoma: a multicentre, open-label, parallel-group, randomised, phase 2 trial. Lancet Oncol. 2020 Apr;21(4):571-580. doi: 10.1016/S1470-2045(20)30011-5. Epub 2020 Feb 26. PMID 32112738
- [Background] Xu J, Shen J, Gu S, Zhang Y, Wu L, Wu J, Shao G, Zhang Y, Xu L, Yin T, Liu J, Ren Z, Xiong J, Mao X, Zhang L, Yang J, Li L, Chen X, Wang Z, Gu K, Chen X, Pan Z, Ma K, Zhou X, Yu Z, Li E, Yin G, Zhang X, Wang S, Wang Q. Camrelizumab in Combination with Apatinib in Patients with Advanced Hepatocellular Carcinoma (RESCUE): A Nonrandomized, Open-label, Phase II Trial. Clin Cancer Res. 2021 Feb 15;27(4):1003-1011. doi: 10.1158/1078-0432.CCR-20-2571. Epub 2020 Oct 21. PMID 33087333
- [Background] Yamamoto Y, Matsui J, Matsushima T, Obaishi H, Miyazaki K, Nakamura K, Tohyama O, Semba T, Yamaguchi A, Hoshi SS, Mimura F, Haneda T, Fukuda Y, Kamata JI, Takahashi K, Matsukura M, Wakabayashi T, Asada M, Nomoto KI, Watanabe T, Dezso Z, Yoshimatsu K, Funahashi Y, Tsuruoka A. Lenvatinib, an angiogenesis inhibitor targeting VEGFR/FGFR, shows broad antitumor activity in human tumor xenograft models associated with microvessel density and pericyte coverage. Vasc Cell. 2014 Sep 6;6:18. doi: 10.1186/2045-824X-6-18. eCollection 2014. PMID 25197551
- [Background] Terme M, Tartour E, Taieb J. VEGFA/VEGFR2-targeted therapies prevent the VEGFA-induced proliferation of regulatory T cells in cancer. Oncoimmunology. 2013 Aug 1;2(8):e25156. doi: 10.4161/onci.25156. Epub 2013 Jun 10. PMID 24083078
- [Background] Hume DA, MacDonald KP. Therapeutic applications of macrophage colony-stimulating factor-1 (CSF-1) and antagonists of CSF-1 receptor (CSF-1R) signaling. Blood. 2012 Feb 23;119(8):1810-20. doi: 10.1182/blood-2011-09-379214. Epub 2011 Dec 20. PMID 22186992
- [Background] Hoff S, Grünewald S, Röse L, Zopf D. 1198PImmunomodulation by regorafenib alone and in combination with anti PD1 antibody on murine models of colorectal cancer. Ann Oncol 2017;28.
- [Background] Shigeta K, Matsui A, Kikuchi H, Klein S, Mamessier E, Chen IX, Aoki S, Kitahara S, Inoue K, Shigeta A, Hato T, Ramjiawan RR, Staiculescu D, Zopf D, Fiebig L, Hobbs GS, Quaas A, Dima S, Popescu I, Huang P, Munn LL, Cobbold M, Goyal L, Zhu AX, Jain RK, Duda DG. Regorafenib combined with PD1 blockade increases CD8 T-cell infiltration by inducing CXCL10 expression in hepatocellular carcinoma. J Immunother Cancer. 2020 Nov;8(2):e001435. doi: 10.1136/jitc-2020-001435. PMID 33234602
- [Background] Sprinzl MF, Galle PR. Current progress in immunotherapy of hepatocellular carcinoma. J Hepatol. 2017 Mar;66(3):482-484. doi: 10.1016/j.jhep.2016.12.009. Epub 2016 Dec 21. No abstract available. PMID 28011330
- [Background] Topalian SL, Drake CG, Pardoll DM. Immune checkpoint blockade: a common denominator approach to cancer therapy. Cancer Cell. 2015 Apr 13;27(4):450-61. doi: 10.1016/j.ccell.2015.03.001. Epub 2015 Apr 6. PMID 25858804
- [Background] Rotte A, Jin JY, Lemaire V. Mechanistic overview of immune checkpoints to support the rational design of their combinations in cancer immunotherapy. Ann Oncol. 2018 Jan 1;29(1):71-83. doi: 10.1093/annonc/mdx686. PMID 29069302
- [Background] Jia Y, Zeng Z, Li Y, Li Z, Jin L, Zhang Z, Wang L, Wang FS. Impaired function of CD4+ T follicular helper (Tfh) cells associated with hepatocellular carcinoma progression. PLoS One. 2015 Feb 17;10(2):e0117458. doi: 10.1371/journal.pone.0117458. eCollection 2015. PMID 25689070
- [Background] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640